CLINICAL TRIAL: NCT01443403
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of S-297995 for the Treatment of Opioid-Induced Constipation in Subjects With Non-Malignant Chronic Pain Receiving Opioid Therapy
Brief Title: A Study of Naldemedine (S-297995) for the Treatment of Opioid-Induced Constipation in Adults With Non-Malignant Chronic Pain Receiving Opioid Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1107V9221
Record Dates: First submitted 2011-09-20; First posted 2011-09-29 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-05

CONDITIONS: Opioid-induced Constipation
Keywords: Opioid Therapy; Non-Malignant Chronic Pain; Opioid-Induced Constipation
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naldemedine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo orally once daily for 28 days.
  Interventions: Drug: Placebo
- Naldemedine 0.1 mg (Experimental): Participants received 0.1 mg naldemedine orally once daily for 28 days.
  Interventions: Drug: Naldemedine
- Naldemedine 0.2 mg (Experimental): Participants received 0.2 mg naldemedine orally once daily for 28 days.
  Interventions: Drug: Naldemedine
- Naldemedine 0.4 mg (Experimental): Participants received 0.4 mg naldemedine orally once daily for 28 days.
  Interventions: Drug: Naldemedine

INTERVENTIONS:
Drug: Placebo — Matching placebo tablets administered orally once a day.
  Arms: Placebo
Drug: Naldemedine — Naldemedine tablets administered orally once a day.
  Other Names: S 297995; Symproic®
  Arms: Naldemedine 0.1 mg; Naldemedine 0.2 mg; Naldemedine 0.4 mg

SUMMARY:
The purpose of this study is to determine efficacy and safety of naldemedine for the treatment of opioid-induced constipation in adults with non-malignant chronic pain receiving opioid therapy for ≥ 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years or older at time of informed consent with non-malignant chronic pain experiencing opioid-induced constipation
* Subjects with < 3 spontaneous bowel movements a week and experiencing bowel symptoms
* Subjects receiving chronic opioid therapy due to non-malignant pain for ≥ 3 months

Exclusion Criteria:

* Evidence of clinically significant gastrointestinal disease
* History of chronic constipation prior to starting analgesic medication or any potential non-opioid cause of bowel dysfunction that may be a major contributor to the constipation
* Severe constipation that has not been appropriately managed such that the subject is at immediate risk of developing serious complications of constipation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2011-08-17 (Actual); Primary Completion 2012-08-22 (Actual); Study Completion 2012-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (49):
- United States (49):
  - Shionogi Research Site, Phoenix, Arizona
  - Shionogi Research Site, Sun Lakes, Arizona
  - Shionogi Research Site, Little Rock, Arkansas
  - Shionogi Research Site, Anaheim, California
  - Shionogi Research Site, Fresno, California
  - Shionogi Research Site, Lincoln, California
  - Shionogi Research Site, Lomita, California
  - Shionogi Research Site, Denver, Colorado
  - Shionogi Research Site, Brandon, Florida
  - Shionogi Research Site, Kissimmee, Florida
  - Shionogi Research Site, New Port Richey, Florida
  - Shionogi Research Site, North Miami, Florida
  - Shionogi Research Site, Ocala, Florida
  - Shionogi Research Site, Orlando, Florida
  - Shionogi Research Site, Ormond Beach, Florida
  - Shionogi Research Site, Port Orange, Florida
  - Shionogi Research Site, Sarasota, Florida
  - Shionogi Research Site, South Miami, Florida
  - Shionogi Research Site, West Palm Beach, Florida
  - Shionogi Research Site, Atlanta, Georgia
  - Shionogi Research Site, Decatur, Georgia
  - Shionogi Research Site, Marietta, Georgia
  - Shionogi Research Site, Evansville, Indiana
  - Shionogi Research Site, Lexington, Kentucky
  - Shionogi Research Site, Shreveport, Louisiana
  - Shionogi Research Site, Owings Mills, Maryland
  - Shionogi Research Site, Watertown, Massachusetts
  - Shionogi Research Site, Worcester, Massachusetts
  - Shionogi Research Site, Traverse City, Michigan
  - Shionogi Research Site, Edina, Minnesota
  - Shionogi Research Site, Las Vegas, Nevada
  - Shionogi Research Site, Newington, New Hampshire
  - Shionogi Research Site, Berlin, New Jersey
  - Shionogi Research Site, Willingboro, New Jersey
  - Shionogi Research Site, Hartsdale, New York
  - Shionogi Research Site, North Syracuse, New York
  - Shionogi Research Site, Williamsville, New York
  - Shionogi Research Site, Wilmington, North Carolina
  - Shionogi Research Site, Winston-Salem, North Carolina
  - Shionogi Research Site, Canton, Ohio
  - Shionogi Research Site, Columbus, Ohio
  - Shionogi Research Site, Perrysburg, Ohio
  - Shionogi Research Site, Eugene, Oregon
  - Shionogi Research Site, Philadelphia, Pennsylvania
  - Shionogi Research Site, Greer, South Carolina
  - Shionogi Research Site, Austin, Texas
  - Shionogi Research Site, Dallas, Texas
  - Shionogi Research Site, Orem, Utah
  - Shionogi Research Site, Salt Lake City, Utah

REFERENCES:
- [Result] Webster LR, Yamada T, Arjona Ferreira JC. A Phase 2b, Randomized, Double-Blind Placebo-Controlled Study to Evaluate the Efficacy and Safety of Naldemedine for the Treatment of Opioid-Induced Constipation in Patients with Chronic Noncancer Pain. Pain Med. 2017 Dec 1;18(12):2350-2360. doi: 10.1093/pm/pnw325. PMID 28371937

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 53 clinical sites in the United States. The first participant was enrolled on August 17, 2011 and the last participant completed on August 22, 2012.
  Participants must have met eligibility criteria and completed the Bowel Movement and Constipation Assessment (BMCA) Diary for a minimum of 14 days to enroll in the study.
Pre-assignment Details: Participants were randomized in a 1:1:1:1 ratio to receive placebo, naldemedine 0.1 mg, 0.2 mg, or 0.4 mg once daily.
  One participant was randomized twice, first to placebo and subsequently to naldemedine 0.4 mg, and is counted in both arms below and for safety analyses.
Period: Overall Study
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Started | 61 | 61 | 61 | 61
Received Treatment | 61 | 61 | 60 | 61
Completed | 55 | 55 | 54 | 52
Not Completed | 6 | 6 | 7 | 9
Not completed — Adverse Event | 1 | 1 | 4 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 1 | 1 | 1
Not completed — Use of Prohibited Treatment | 2 | 3 | 0 | 0
Not completed — Other - Miscellaneous | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The modified intention-to-treat (mITT) population included all randomized participants who received study drug and had at least 1 postdose primary efficacy assessment completed. One participant who randomized twice was excluded from the naldemedine 0.4 mg arm for the mITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg | Total
Number analyzed (Participants) | 61 | 61 | 59 | 57 | 238
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.1 (10.88) | 49.5 (9.71) | 50.7 (11.40) | 54.1 (11.19) | 51.9 (10.80)
Age, Customized [Number; unit: participants]
  ≥ 18 - < 40 years | 6 | 10 | 13 | 7 | 36
  ≥ 40 - < 50 years | 14 | 18 | 8 | 12 | 52
  ≥ 50 - < 65 years | 33 | 31 | 34 | 29 | 127
  ≥ 65 - < 75 years | 6 | 2 | 3 | 8 | 19
  ≥ 75 years | 2 | 0 | 1 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 47 | 38 | 37 | 167
  Male | 16 | 14 | 21 | 20 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 2 | 4 | 16
  Not Hispanic or Latino | 57 | 55 | 57 | 53 | 222
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Naive | 2 | 0 | 0 | 0 | 2
  Asian | 1 | 0 | 0 | 0 | 1
  Black or African American | 9 | 11 | 12 | 6 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 49 | 49 | 47 | 51 | 196
  Other | 0 | 1 | 0 | 0 | 1
Spontaneous Bowel Movement (SBM) Frequency per Week [Mean (Standard Deviation); unit: SBMs/week] | 1.22 (0.720) | 1.51 (0.820) | 1.52 (0.916) | 1.20 (0.948) | 1.36 (0.851)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Last 2 Weeks of the Treatment Period in the Number of Spontaneous Bowel Movements Per Week
Description: Participants completed a daily Bowel Movement and Constipation Assessment Diary to record information about bowel movements and constipation.
  A spontaneous bowel movement was defined as a bowel movement unassisted by rescue medication (laxative or enema) taken within the 24 hours preceding the bowel movement. Baseline was defined as the average number of SBMs per week during the 2 weeks prior to randomization. The number of SBMs per week in the last 2 weeks of treatment is defined as the average number of SBMs per week recorded in the diary for the 14 days prior to the last dose of study drug.
Time Frame: Baseline (2 weeks prior to randomization) and the last 2 weeks of treatment (Weeks 3 to 4 for participants who completed the 28-day treatment period)
Population: Modified intention-to-treat population
Measure: Least Squares Mean (Standard Error); unit: spontaneous bowel movements per week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
spontaneous bowel movements per week | 1.42 (0.422) | 1.98 (0.422) | 3.37 (0.429) | 3.64 (0.437)
Statistical Analysis 1: Comparison: Placebo vs Naldemedine 0.4 mg; Test type: Superiority or Other; p = 0.0003, ANCOVA; Analysis of covariance (ANCOVA) model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 2.22, 95% CI 2-sided [1.02 to 3.41], Standard Error of Mean 0.605
Statistical Analysis 2: Comparison: Placebo vs Naldemedine 0.2 mg; Test type: Superiority or Other; p = 0.0014, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 1.95, 95% CI 2-sided [0.76 to 3.14], Standard Error of Mean 0.604
Statistical Analysis 3: Comparison: Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.3504, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 0.56, 95% CI 2-sided [-0.62 to 1.74], Standard Error of Mean 0.599

2. Secondary Outcome: Change From Baseline to Weeks 1, 2, 3, and 4 in the Number of Spontaneous Bowel Movements Per Week
Description: Participants completed a daily Bowel Movement and Constipation Assessment Diary to record information about bowel movements and constipation.
  A spontaneous bowel movement was defined as a bowel movement unassisted by rescue medication (laxative or enema) taken within the 24 hours preceding the bowel movement. Baseline was defined as the average number of SBMs per day during the 2 weeks prior to randomization.
Time Frame: Baseline and Weeks 1, 2, 3, and 4
Population: mITT population with values at both baseline and the specified time point.
Measure: Least Squares Mean (Standard Error); unit: spontaneous bowel movements per week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
spontaneous bowel movements per week
  Week 1 (n = 61, 61, 59, 57) | 1.61 (0.507) | 2.21 (0.507) | 4.05 (0.516) | 4.52 (0.525)
  Week 2 (n = 61, 60, 59, 56) | 1.53 (0.402) | 2.06 (0.402) | 2.99 (0.410) | 3.87 (0.416)
  Week 3 (n = 60, 60, 59, 57) | 1.32 (0.374) | 2.27 (0.372) | 3.07 (0.380) | 3.33 (0.384)
  Week 4 (n = 60, 60, 59, 57) | 1.36 (0.409) | 1.69 (0.409) | 3.30 (0.415) | 3.41 (0.420)

3. Secondary Outcome: Change From Baseline to the Last 2 Weeks of the Treatment Period in the Number of Bowel Movements (BMs) Per Week
Description: Participants completed a daily Bowel Movement and Constipation Assessment Diary to record information about bowel movements and constipation.
  A BM was defined as all bowel movements observed irrespective of the use of a laxative agent.
Time Frame: Baseline and the last 2 weeks of treatment (Weeks 3 to 4 for participants who completed the 28-day treatment period)
Population: mITT population
Measure: Least Squares Mean (Standard Error); unit: bowel movements per week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
bowel movements per week | 1.43 (0.396) | 2.07 (0.394) | 3.35 (0.404) | 3.36 (0.408)
Statistical Analysis 1: Comparison: Placebo vs Naldemedine 0.4 mg; Test type: Superiority or Other; p = 0.0008, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 1.93, 95% CI 2-sided [0.81 to 3.05], Standard Error of Mean 0.568
Statistical Analysis 2: Comparison: Placebo vs Naldemedine 0.2 mg; Test type: Superiority or Other; p = 0.0009, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 1.91, 95% CI 2-sided [0.79 to 3.04], Standard Error of Mean 0.569
Statistical Analysis 3: Comparison: Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.2572, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 0.63, 95% CI 2-sided [-0.47 to 1.73], Standard Error of Mean 0.558

4. Secondary Outcome: Change From Baseline to Weeks 1, 2, 3, and 4 in the Number of Bowel Movements Per Week
Description: as for outcome 3
Time Frame: Baseline and Weeks 1, 2, 3, and 4
Population: mITT population with values at both baseline and the specified time point.
Measure: Least Squares Mean (Standard Error); unit: bowel movements per week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
bowel movements per week
  Week 1 (n = 61, 61, 59, 57) | 1.67 (0.457) | 2.27 (0.456) | 4.25 (0.466) | 4.60 (0.472)
  Week 2 (n = 61, 60, 59, 56) | 1.65 (0.361) | 1.97 (0.360) | 2.96 (0.369) | 3.75 (0.373)
  Week 3 (n = 60, 60, 59, 57) | 1.36 (0.347) | 2.36 (0.344) | 3.02 (0.352) | 2.93 (0.354)
  Week 4 (n = 60, 60, 59, 57) | 1.52 (0.373) | 1.68 (0.372) | 3.06 (0.379) | 3.16 (0.381)

5. Secondary Outcome: Change From Baseline to the Last 2 Weeks of the Treatment Period in the Number of Complete Bowel Movements (CBMs) Per Week
Description: Participants completed a daily Bowel Movement and Constipation Assessment Diary to record information about bowel movements and constipation.
  A complete BM (CBM) was defined as a BM where the participant answered 'Yes' to the following question: 'Did you have a feeling of complete emptying after the bowel movement?'
Time Frame: Baseline and the last 2 weeks of treatment (Weeks 3 to 4 for participants who completed the 28-day treatment period)
Population: mITT population
Measure: Least Squares Mean (Standard Error); unit: complete bowel movements per week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
complete bowel movements per week | 1.08 (0.336) | 1.58 (0.336) | 2.71 (0.344) | 2.41 (0.348)
Statistical Analysis 1: Comparison: Placebo vs Naldemedine 0.4 mg; Test type: Superiority or Other; p = 0.0065, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 1.33, 95% CI 2-sided [0.38 to 2.28], Standard Error of Mean 0.484
Statistical Analysis 2: Comparison: Placebo vs Naldemedine 0.2 mg; Test type: Superiority or Other; p = 0.0008, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 1.64, 95% CI 2-sided [0.69 to 2.58], Standard Error of Mean 0.482
Statistical Analysis 3: Comparison: Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.2921, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 0.50, 95% CI 2-sided [-0.43 to 1.44], Standard Error of Mean 0.476

6. Secondary Outcome: Change From Baseline to Weeks 1, 2, 3, and 4 in the Number of Complete Bowel Movements Per Week
Description: as for outcome 5
Time Frame: Baseline and Weeks 1, 2, 3, and 4
Population: mITT population with values at both baseline and the specified time point.
Measure: Least Squares Mean (Standard Error); unit: complete bowel movements per week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
complete bowel movements per week
  Week 1 (n = 61, 61, 59, 57) | 0.73 (0.381) | 1.38 (0.380) | 2.88 (0.388) | 3.14 (0.394)
  Week 2 (n = 61, 60, 59, 56) | 1.07 (0.324) | 1.54 (0.324) | 1.99 (0.331) | 2.50 (0.336)
  Week 3 (n = 60, 60, 59, 57) | 1.11 (0.297) | 1.62 (0.296) | 2.29 (0.302) | 2.12 (0.305)
  Week 4 (n = 60, 60, 59, 57) | 1.09 (0.334) | 1.60 (0.333) | 2.77 (0.339) | 2.56 (0.342)

7. Secondary Outcome: Change From Baseline to the Last 2 Weeks of the Treatment Period in the Number of Complete Spontaneous Bowel Movements (CSBMs) Per Week
Description: Participants completed a daily Bowel Movement and Constipation Assessment Diary to record information about bowel movements and constipation.
  A CSBM was defined as a spontaneous BM which was accompanied by the feeling of complete evacuation.
Time Frame: Baseline and the last 2 weeks of treatment (Weeks 3 to 4 for participants who completed the 28-day treatment period)
Population: mITT population
Measure: Least Squares Mean (Standard Error); unit: complete spontaneous BMs per week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
complete spontaneous BMs per week | 0.99 (0.345) | 1.49 (0.344) | 2.69 (0.351) | 2.44 (0.356)
Statistical Analysis 1: Comparison: Placebo vs Naldemedine 0.4 mg; Test type: Superiority or Other; p = 0.0039, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 1.44, 95% CI 2-sided [0.47 to 2.42], Standard Error of Mean 0.495
Statistical Analysis 2: Comparison: Placebo vs Naldemedine 0.2 mg; Test type: Superiority or Other; p = 0.0007, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 1.70, 95% CI 2-sided [0.73 to 2.67], Standard Error of Mean 0.492
Statistical Analysis 3: Comparison: Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.3077, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 0.50, 95% CI 2-sided [-0.46 to 1.46], Standard Error of Mean 0.488

8. Secondary Outcome: Change From Baseline to Weeks 1, 2, 3, and 4 in the Number of Complete Spontaneous Bowel Movements Per Week
Description: as for outcome 7
Time Frame: Baseline and Weeks 1, 2, 3, and 4
Population: mITT population with values at both baseline and the specified time point.
Measure: Least Squares Mean (Standard Error); unit: complete spontaneous BMs per week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
complete spontaneous BMs per week
  Week 1 (n = 61, 61, 59, 57) | 0.71 (0.386) | 1.31 (0.386) | 2.63 (0.393) | 2.99 (0.399)
  Week 2 (n = 61, 60, 59, 56) | 1.09 (0.326) | 1.41 (0.326) | 2.08 (0.332) | 2.50 (0.337)
  Week 3 (n = 60, 60, 59, 57) | 1.02 (0.303) | 1.53 (0.301) | 2.28 (0.307) | 2.21 (0.311)
  Week 4 (n = 60, 60, 59, 57) | 0.90 (0.340) | 1.51 (0.340) | 2.77 (0.345) | 2.58 (0.349)

9. Secondary Outcome: Percentage of Participants With an SBM Response in the Last 2 Weeks of the Treatment Period
Description: Participants completed a daily Bowel Movement and Constipation Assessment Diary to record information about bowel movements and constipation.
  An SBM responder was defined as a participant whose frequency of SBMs within the last 2 weeks of the treatment period was 3 times or more per week and who had an average increase in the frequency of SBMs from baseline of 1 or more per week.
Time Frame: Baseline and the last 2 weeks of treatment (Weeks 3 to 4 for participants who completed the 28-day treatment period)
Population: mITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
percentage of participants | 39.3 | 52.5 | 71.2 | 66.7
Statistical Analysis 1: Comparison: Placebo vs Naldemedine 0.4 mg; Test type: Superiority or Other; p = 0.0030, Chi-squared; Difference = 27.3, 95% CI 2-sided [10.0 to 44.6]
Statistical Analysis 2: Comparison: Placebo vs Naldemedine 0.2 mg; Test type: Superiority or Other; p = 0.0005, Chi-squared; Difference = 31.8, 95% CI 2-sided [15.0 to 48.7]
Statistical Analysis 3: Comparison: Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.1461, Chi-squared; Difference = 13.1, 95% CI 2-sided [-4.4 to 30.6]

10. Secondary Outcome: Percentage of Participants With an SBM Response at Weeks 1, 2, 3 and 4
Description: Participants completed a daily Bowel Movement and Constipation Assessment Diary to record information about bowel movements and constipation.
  An SBM responder was defined as any participant whose frequency of SBM per week during the treatment period was 3 times or more per week, and who had an average increase from baseline of 1 or more per week.
Time Frame: Baseline and Weeks 1, 2, 3, and 4
Population: mITT population; missing data were imputed using last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
percentage of participants
  Week1 | 45.9 | 62.3 | 72.9 | 70.2
  Week 2 | 45.9 | 55.7 | 69.5 | 70.2
  Week 3 | 45.9 | 55.7 | 74.6 | 73.7
  Week 4 | 39.3 | 42.6 | 64.4 | 64.9

11. Secondary Outcome: Percentage of Participants With a CSBM Response in the Last 2 Weeks of the Treatment Period
Description: Participants completed a daily Bowel Movement and Constipation Assessment Diary to record information about bowel movements and constipation.
  A CSBM responder was defined as a participant whose frequency of CSBMs within the last 2 weeks of the treatment period was 3 times or more per week and who had an average increase in the frequency of CSBMs from baseline of 1 or more per week.
Time Frame: Baseline and the last 2 weeks of treatment (Weeks 3 to 4 for participants who completed the 28-day treatment period)
Population: mITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
percentage of participants | 21.3 | 29.5 | 45.8 | 45.6
Statistical Analysis 1: Comparison: Placebo vs Naldemedine 0.4 mg; Test type: Superiority or Other; p = 0.0050, Chi-squared; Difference = 24.3, 95% CI 2-sided [7.8 to 40.8]
Statistical Analysis 2: Comparison: Placebo vs Naldemedine 0.2 mg; Test type: Superiority or Other; p = 0.0045, Chi-squared; Difference = 24.5, 95% CI 2-sided [8.1 to 40.8]
Statistical Analysis 3: Comparison: Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.2984, Chi-squared; Difference = 8.2, 95% CI 2-sided [-7.2 to 23.6]

12. Secondary Outcome: Percentage of Participants With a CSBM Response at Weeks 1, 2, 3, and 4
Description: Participants completed a daily Bowel Movement and Constipation Assessment Diary to record information about bowel movements and constipation.
  A CSBM responder was defined as a participant whose frequency of CSBMs during the treatment period was 3 times or more per week and who had an average increase in the frequency of CSBMs from baseline of 1 or more per week.
Time Frame: Baseline and Weeks 1, 2, 3, and 4
Population: mITT population; missing data were imputed using last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
percentage of participants
  Week 1 | 21.3 | 31.1 | 42.4 | 50.9
  Week 2 | 23.0 | 29.5 | 42.4 | 40.4
  Week 3 | 24.6 | 37.7 | 44.1 | 45.6
  Week 4 | 21.3 | 27.9 | 45.8 | 43.9

13. Secondary Outcome: Change From Baseline to the Last 2 Weeks of the Treatment Period in Number of Days Per Week With SBMs
Description: Participants completed a daily Bowel Movement and Constipation Assessment Diary to record information about bowel movements and constipation.
  An SBM is defined as a bowel movement unassisted by rescue medication (laxative or enema) taken within the 24 hours preceding the bowel movement.
Time Frame: Baseline and the last 2 weeks of treatment (Weeks 3 to 4 for participants who completed the 28-day treatment period)
Population: mITT population
Measure: Least Squares Mean (Standard Error); unit: days/week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
days/week | 0.88 (0.223) | 1.46 (0.223) | 2.10 (0.227) | 2.42 (0.232)
Statistical Analysis 1: Comparison: Placebo vs Naldemedine 0.4 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 1.54, 95% CI 2-sided [0.90 to 2.17], Standard Error of Mean 0.320
Statistical Analysis 2: Comparison: Placebo vs Naldemedine 0.2 mg; Test type: Superiority or Other; p = 0.0002, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 1.22, 95% CI 2-sided [0.59 to 1.85], Standard Error of Mean 0.320
Statistical Analysis 3: Comparison: Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.0698, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 0.58, 95% CI 2-sided [-0.05 to 1.20], Standard Error of Mean 0.317

14. Secondary Outcome: Change From Baseline to Weeks 1, 2, 3 and 4 in Number of Days Per Week With SBMs
Description: as for outcome 13
Time Frame: Baseline and Weeks 1, 2, 3, and 4
Population: mITT population with values at both baseline and the specified time point.
Measure: Least Squares Mean (Standard Error); unit: days/week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
days/week
  Week 1 (n = 61, 61, 59, 57) | 1.12 (0.250) | 1.62 (0.251) | 2.35 (0.255) | 2.38 (0.260)
  Week 2 (n = 61, 60, 59, 56) | 1.03 (0.240) | 1.56 (0.240) | 2.03 (0.245) | 2.45 (0.250)
  Week 3 (n = 60, 60, 59, 57) | 0.89 (0.233) | 1.57 (0.232) | 2.07 (0.237) | 2.37 (0.240)
  Week 4 (n = 60, 60, 59, 57) | 0.75 (0.274) | 1.27 (0.274) | 2.20 (0.278) | 2.52 (0.281)

15. Secondary Outcome: Change From Baseline to the Last 2 Weeks of the Treatment Period in Number of Days Per Week With CSBMs
Description: as for outcome 7
Time Frame: Baseline and the last 2 weeks of treatment (Weeks 3 to 4 for participants who completed the 28-day treatment period)
Population: mITT population
Measure: Least Squares Mean (Standard Error); unit: days/week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
days/week | 0.83 (0.214) | 1.25 (0.213) | 1.93 (0.217) | 2.02 (0.221)
Statistical Analysis 1: Comparison: Placebo vs Naldemedine 0.4 mg; Test type: Superiority or Other; p = 0.0001, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 1.19, 95% CI 2-sided [0.58 to 1.79], Standard Error of Mean 0.307
Statistical Analysis 2: Comparison: Placebo vs Naldemedine 0.2 mg; Test type: Superiority or Other; p = 0.0004, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 1.10, 95% CI 2-sided [0.49 to 1.70], Standard Error of Mean 0.305
Statistical Analysis 3: Comparison: Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.1648, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 0.42, 95% CI 2-sided [-0.17 to 1.02], Standard Error of Mean 0.302

16. Secondary Outcome: Change From Baseline to Weeks 1, 2, 3 and 4 in Number of Days Per Week With CSBMs
Description: as for outcome 7
Time Frame: Baseline and Weeks 1, 2, 3, and 4
Population: mITT population with values at both baseline and the specified time point.
Measure: Least Squares Mean (Standard Error); unit: days/week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
days/week
  Week 1 (n = 61, 61, 59, 57) | 0.65 (0.234) | 1.17 (0.234) | 1.74 (0.238) | 2.14 (0.242)
  Week 2 (n = 61, 60, 59, 56) | 0.90 (0.226) | 1.18 (0.226) | 1.65 (0.230) | 1.93 (0.234)
  Week 3 (n = 60, 60, 59, 57) | 0.86 (0.224) | 1.26 (0.223) | 1.71 (0.228) | 1.98 (0.230)
  Week 4 (n = 60, 60, 59, 57) | 0.71 (0.256) | 1.31 (0.256) | 2.17 (0.260) | 2.10 (0.262)

17. Secondary Outcome: Time to the First Spontaneous Bowel Movement
Description: Time to the first SBM was defined as the time to the first SBM after the initial administration of study drug. Participants who withdrew from the study before an SBM was observed or had no SBM during the treatment period were treated as censored.
Time Frame: 28 days
Population: mITT population
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
hours | 49.57 [34.70 to 71.25] | 28.15 [15.75 to 45.02] | 11.08 [4.15 to 25.25] | 21.33 [4.67 to 26.92]
Statistical Analysis 1: Comparison: Placebo vs Naldemedine 0.4 mg; Test type: Superiority or Other; p = 0.0004, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Naldemedine 0.2 mg; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.0118, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Time to the First Complete Spontaneous Bowel Movement
Description: Time to the first CSBM was defined as the time to the first CSBM after the initial administration of study drug. Participants who withdrew from the study before a CSBM was observed or had no CSBM during the treatment period were treated as censored.
Time Frame: 28 days
Population: mITT population
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
hours | 223.92 [101.25 to 350.40] | 82.50 [49.30 to 140.40] | 44.83 [25.58 to 107.17] | 32.93 [18.00 to 55.08]
Statistical Analysis 1: Comparison: Placebo vs Naldemedine 0.4 mg; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Naldemedine 0.2 mg; Test type: Superiority or Other; p = 0.0011, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.0079, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Percentage of Participants With SBMs Within 4, 8, 12, and 24 Hours After the Initial Administration of Study Drug
Description: The percentage of participants who experienced at least one SBM within 4, 8, 12, and 24 hours after the initial administration of study drug and before the second administration.
Time Frame: 4, 8, 12, and 24 hours
Population: mITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
percentage of participants
  Up to 4 hours | 8.2 | 18.0 | 35.6 | 31.6
  Up to 8 hours | 16.4 | 29.5 | 47.5 | 42.1
  Up to 12 hours | 18.0 | 34.4 | 50.8 | 43.9
  Up to 24 hours | 27.9 | 44.3 | 59.3 | 59.6

20. Secondary Outcome: Percentage of Participants With CSBMs Within 4, 8, 12, and 24 Hours After the Initial Administration of Study Drug
Description: The percentage of participants who experienced at least one CSBM within 4, 8, 12, and 24 hours after the initial administration of study drug and before the second administration.
Time Frame: 4, 8, 12, and 24 hours
Population: mITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
percentage of participants
  Up to 4 hours | 1.6 | 11.5 | 18.6 | 12.3
  Up to 8 hours | 6.6 | 16.4 | 20.3 | 24.6
  Up to 12 hours | 6.6 | 21.3 | 23.7 | 33.3
  Up to 24 hours | 14.8 | 27.9 | 30.5 | 43.9

21. Secondary Outcome: Change From Baseline to the Last 2 Weeks of the Treatment Period in Number of SBMs Per Week Rated as 3 or 4 on the Bristol Stool Scale
Description: Consistency of BMs was measured using the Bristol Stool Scale, according to the following: 1 = separate hard lumps like nuts; 2 = sausage shaped but lumpy; 3 = like a sausage, but with cracks on its surface; 4 = like a sausage or a snake, smooth and soft; 5 = soft blobs and with clear-cut edges; 6 = floppy pieces with ragged edges/mushy stool; 7 = watery, no solid pieces, entirely liquid.
Time Frame: Baseline and the last 2 weeks of treatment (Weeks 3 to 4 for participants who completed the 28-day treatment period)
Population: mITT population
Measure: Least Squares Mean (Standard Error); unit: spontaneous bowel movements/week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
spontaneous bowel movements/week | 0.54 (0.249) | 1.08 (0.249) | 2.05 (0.256) | 1.87 (0.259)
Statistical Analysis 1: Comparison: Placebo vs Naldemedine 0.4 mg; Test type: Superiority or Other; p = 0.0003, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 1.33, 95% CI 2-sided [0.62 to 2.03], Standard Error of Mean 0.358
Statistical Analysis 2: Comparison: Placebo vs Naldemedine 0.2 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 1.51, 95% CI 2-sided [0.80 to 2.22], Standard Error of Mean 0.359
Statistical Analysis 3: Comparison: Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.1211, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 0.55, 95% CI 2-sided [-0.15 to 1.24], Standard Error of Mean 0.352

22. Secondary Outcome: Change From Baseline to Weeks 1, 2, 3, and 4 in Number of SBMs Rated as 3 or 4 on the Bristol Stool Scale Per Week
Description: as for outcome 21
Time Frame: Baseline and Weeks 1, 2, 3, and 4
Population: mITT population with values at both baseline and the specified time point.
Measure: Least Squares Mean (Standard Error); unit: spontaneous bowel movements/week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
spontaneous bowel movements/week
  Week 1 (n = 61, 61, 59, 57) | 0.60 (0.278) | 0.97 (0.278) | 2.16 (0.285) | 1.76 (0.288)
  Week 2 (n = 61, 60, 59, 56) | 0.62 (0.271) | 1.19 (0.270) | 2.03 (0.278) | 1.98 (0.281)
  Week 3 (n = 60, 60, 59, 57) | 0.58 (0.262) | 1.08 (0.261) | 2.03 (0.268) | 1.91 (0.270)
  Week 4 (n = 60, 60, 59, 57) | 0.50 (0.307) | 1.10 (0.307) | 2.01 (0.313) | 1.94 (0.315)

23. Secondary Outcome: Change From Baseline to the Last 2 Weeks of the Treatment Period in Number of SBMs Per Week With no Straining
Description: Straining during BMs was graded using the following scale: 0 = No straining; 1 = Mild straining; 2 = Moderate; 3 = Severe; 4 = Very Severe. A BM without straining was defined as a BM with a straining score of 0 or 1.
Time Frame: Baseline and the last 2 weeks of treatment (Weeks 3 to 4 for participants who completed the 28-day treatment period)
Population: mITT population
Measure: Least Squares Mean (Standard Error); unit: bowel movements/week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
bowel movements/week | 0.85 (0.384) | 1.54 (0.383) | 2.92 (0.391) | 3.21 (0.396)
Statistical Analysis 1: Comparison: Placebo vs Naldemedine 0.4 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 2.36, 95% CI 2-sided [1.28 to 3.45], Standard Error of Mean 0.551
Statistical Analysis 2: Comparison: Placebo vs Naldemedine 0.2 mg; Test type: Superiority or Other; p = 0.0002, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 2.07, 95% CI 2-sided [0.99 to 3.15], Standard Error of Mean 0.549
Statistical Analysis 3: Comparison: Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.2022, ANCOVA; ANCOVA model with treatment group as a term and baseline value as a covariate; LS Mean Difference = 0.69, 95% CI 2-sided [-0.37 to 1.76], Standard Error of Mean 0.542

24. Secondary Outcome: Change From Baseline to Weeks 1, 2, 3, and 4 in the Number of SBMs Per Week Without Straining
Description: Straining during BMs was graded using the following scale: 0 = No straining; 1 = Mild straining; 2 = Moderate; 3 = Severe; 4 = Very Severe. A BM without straining is defined as a BM with a straining score of 0 or 1.
Time Frame: Baseline and Weeks 1, 2, 3, and 4
Population: mITT population with values at both baseline and the specified time point.
Measure: Least Squares Mean (Standard Error); unit: bowel movements/week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
bowel movements/week
  Week 1 (n = 61, 61, 59, 57) | 0.97 (0.443) | 1.42 (0.442) | 3.23 (0.451) | 3.46 (0.457)
  Week 2 (n = 61, 60, 59, 56) | 0.97 (0.382) | 1.43 (0.382) | 2.54 (0.390) | 3.27 (0.394)
  Week 3 (n = 60, 60, 59, 57) | 0.94 (0.371) | 1.70 (0.369) | 2.67 (0.377) | 3.06 (0.381)
  Week 4 (n = 60, 60, 59, 57) | 0.61 (0.359) | 1.39 (0.358) | 2.82 (0.365) | 2.84 (0.368)

25. Secondary Outcome: Change From Baseline to the Last 2 Weeks of the Treatment Period in Number of False Start BMs Per Week
Description: Participants completed a daily Bowel Movement and Constipation Assessment Diary to record information about bowel movements and constipation.
  A false start was defined as any attempted, but unsuccessful bowel movement (no solid or liquid fecal material was excreted).
Time Frame: Baseline and the last 2 weeks of treatment (Weeks 3 to 4 for participants who completed the 28-day treatment period)
Population: mITT population with values at both baseline and the last 2 weeks of the treatment period
Measure: Mean (Standard Deviation); unit: false start BMs
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 60 | 61 | 58 | 57
false start BMs | -2.71 (5.105) | -3.06 (4.568) | -3.75 (5.673) | -2.80 (5.353)

26. Secondary Outcome: Change From Baseline to the Last 2 Weeks of the Treatment Period in Rescue Use of Laxative Agents Per Week
Description: Participants were asked how many doses of rescue laxative medication they had taken within the past 24 hours as part of the Bowel Movement and Constipation Assessment Diary (BMCA).
Time Frame: Baseline and the last 2 weeks of treatment (Weeks 3 to 4 for participants who completed the 28-day treatment period)
Population: mITT population
Measure: Mean (Standard Deviation); unit: doses/week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
doses/week | 0.94 (6.068) | -0.47 (1.691) | 0.15 (07.211) | -1.24 (2.847)
Statistical Analysis 1: Comparison: Placebo vs Naldemedine 0.4 mg; Test type: Superiority or Other; p = 0.0272, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Naldemedine 0.2 mg; Test type: Superiority or Other; p = 0.1355, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.3689, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Mean Rescue Laxative Use Per Week During the Treatment Period
Description: as for outcome 26
Time Frame: Weeks 1 to 4
Population: mITT population
Measure: Mean (Standard Deviation); unit: doses/week
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
doses/week | 2.9 (6.98) | 0.9 (1.81) | 2.9 (7.64) | 1.8 (4.86)

28. Secondary Outcome: Change From Baseline to the Last 2 Weeks of the Treatment Period in Abdominal Bloating
Description: Participants were asked to rate their abdominal bloating for the past 24 hours on a scale of 0 to 4, where 0 = Absent; 1 = Mild; 2 = Moderate; 3 = Severe; 4 = Very Severe.
Time Frame: Baseline and the last 2 weeks of treatment (Weeks 3 to 4 for participants who completed the 28-day treatment period)
Population: mITT population with a value at both baseline and the last 2 weeks of treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 60 | 61 | 58 | 57
units on a scale | -0.40 (0.689) | -0.46 (0.759) | -0.54 (0.719) | -0.57 (0.773)
Statistical Analysis 1: Comparison: Placebo vs Naldemedine 0.4 mg; Test type: Superiority or Other; p = 0.2126, Welch's t-test
Statistical Analysis 2: Comparison: Placebo vs Naldemedine 0.2 mg; Test type: Superiority or Other; p = 0.2799, Welch's t-test
Statistical Analysis 3: Comparison: Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.6466, Welch's t-test

29. Secondary Outcome: Change From Baseline to Weeks 1, 2, 3, and 4 in Abdominal Bloating
Description: as for outcome 28
Time Frame: Baseline and Weeks 1, 2, 3, and 4
Population: mITT population with a value at both baseline and the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
units on a scale
  Week 1 (n = 61, 61, 59, 57) | -0.20 (0.592) | -0.30 (0.621) | -0.34 (0.760) | -0.48 (0.692)
  Week 2 (n = 61, 61, 59, 56) | -0.36 (0.654) | -0.45 (0.812) | -0.40 (0.839) | -0.68 (0.745)
  Week 3 (n = 61, 61, 59, 57) | -0.33 (0.666) | -0.40 (0.874) | -0.44 (0.933) | -0.57 (0.818)
  Week 4 (n = 61, 61, 59, 57) | -0.41 (0.652) | -0.51 (0.769) | -0.47 (0.903) | -0.63 (0.784)

30. Secondary Outcome: Change From Baseline to the Last 2 Weeks of the Treatment Period in Abdominal Discomfort
Description: Participants were asked to rate their abdominal discomfort for the past 24 hours on a scale from 0 to 4, where 0 = Absent; 1 = Mild; 2 = Moderate; 3 = Severe; 4 = Very Severe.
Time Frame: Baseline and the last 2 weeks of treatment (Weeks 3 to 4 for participants who completed the 28-day treatment period)
Population: mITT population with a value at both baseline and the last 2 weeks of treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 60 | 61 | 58 | 57
units on a scale | -0.42 (0.730) | -0.51 (0.787) | -0.50 (0.703) | -0.42 (0.991)
Statistical Analysis 1: Comparison: Placebo vs Naldemedine 0.4 mg; Test type: Superiority or Other; p = 0.9826, Welch's t-test
Statistical Analysis 2: Comparison: Placebo vs Naldemedine 0.2 mg; Test type: Superiority or Other; p = 0.5188, Welch's t-test
Statistical Analysis 3: Comparison: Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.5029, Welch's t-test

31. Secondary Outcome: Change From Baseline to Weeks 1, 2, 3, and 4 in Abdominal Discomfort
Description: as for outcome 30
Time Frame: Baseline and Weeks 1, 2, 3, and 4
Population: mITT population with a value at both baseline and the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
units on a scale
  Week 1 (n = 61, 61, 59, 57) | -0.22 (0.652) | -0.35 (0.609) | -0.24 (0.755) | -0.23 (0.652)
  Week 2 (n = 61, 61, 59, 56) | -0.27 (0.705) | -0.48 (0.752) | -0.39 (0.825) | -0.49 (0.713)
  Week 3 (n = 61, 61, 59, 57) | -0.36 (0.741) | -0.43 (0.859) | -0.42 (0.884) | -0.45 (1.001)
  Week 4 (n = 61, 61, 59, 57) | -0.40 (0.684) | -0.51 (0.787) | -0.50 (0.703) | -0.42 (0.991)

32. Secondary Outcome: Subject Global Satisfaction at End of Treatment
Description: On day 29 (or at early termination), participants were asked about their degree of satisfaction with constipation and abdominal symptoms from the start of study drug dosing to Day 28 (or early termination visit). The grades were as follows: 1, markedly worsened; 2, moderately worsened; 3, slightly worsened; 4, unchanged; 5, slightly improved; 6, moderately improved; and 7, markedly improved.
Time Frame: Day 29, or at early termination
Population: mITT population
Measure: Number; unit: participants
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 59 | 57
participants
  Markedly worsened | 1 | 0 | 0 | 1
  Moderately worsened | 2 | 2 | 0 | 2
  Slightly worsened | 3 | 2 | 1 | 0
  Unchanged | 23 | 12 | 4 | 6
  Slightly improved | 12 | 18 | 17 | 8
  Moderately improved | 14 | 17 | 21 | 13
  Markedly improved | 3 | 7 | 14 | 23
  Missing | 3 | 3 | 2 | 4

33. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Naldemedine and Metabolite Nor-S-297995
Description: Pharmacokinetic blood samples for naldemedine (S-297995) and its metabolite, Nor-S-297995, were collected from a subset of participants at selected study sites on Day 1 and in a further subset on Day 28.
Time Frame: Day 1 and Day 28 predose and 1, 2, 4, 8, and 24 hours postdose
Population: The PK parameter population (PK population) includes all participants who received study drug with at least one PK parameter estimated adequately on Day 1 or Day 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 9 | 9 | 10
ng/mL
  Naldemedine Day 1 (n = 9, 9, 10) | 0.987 (41.1) | 1.89 (48.2) | 3.67 (41.3)
  Naldemedine Day 28 (n = 4, 4, 4) | 1.15 (25.8) | 2.00 (22.7) | 4.03 (32.3)
  Nor-S-297995 Day 1 (n = 9, 9, 10) | NA (NA) — Not calculable as plasma concentrations of Nor-S-297995 on Day 1 were below the limit of quantification. | 0.107 (7.8) | 0.184 (30.9)
  Nor-S-297995 Day 28 (n = 4, 4, 4) | 0.111 (27.1) | 0.148 (59.9) | 0.218 (58.3)

34. Secondary Outcome: Time to Maximum Concentration (Tmax) of Naldemedine and Metabolite Nor-S-297995
Description: as for outcome 33
Time Frame: Day 1 and Day 28 predose and 1, 2 , 4, 8, and 24 hours postdose
Population: PK population with available data
Measure: Median (Full Range); unit: hours
Arm/Group | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 9 | 9 | 10
hours
  Naldemedine Day 1 (n = 9, 9, 10) | 1.00 [0.97 to 2.27] | 1.03 [0.97 to 4.02] | 1.03 [0.95 to 4.00]
  Naldemedine Day 28 (n = 4, 4, 4) | 1.03 [1.00 to 1.97] | 1.00 [1.00 to 1.03] | 1.00 [1.00 to 1.08]
  Nor-S-297995 Day 1 (n = 9, 5, 9) | NA [NA to NA] — Not calculable as plasma concentrations of Nor-S-297995 on Day 1 were below the limit of quantification. | 4.00 [2.00 to 8.00] | 4.03 [2.00 to 8.00]
  Nor-S-297995 Day 28 (n = 3, 4, 4) | 2.02 [2.00 to 4.00] | 4.00 [3.97 to 8.03] | 3.00 [2.00 to 4.00]

35. Secondary Outcome: Area Under the Concentration-time Curve From Hour 0 to the Time Point of the Last Measurable Concentration Within the Dose Interval (AUC0-τ)
Description: as for outcome 33
Time Frame: Day 1 and Day 28 predose and 1, 2 , 4, 8, and 24 hours postdose
Population: PK population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 9 | 9 | 10
ng*hr/mL
  Naldemedine Day 1 (n = 6, 8, 7) | 8.491 (24.5) | 15.95 (42.6) | 30.58 (26.9)
  Naldemedine Day 28 (n = 3, 4, 3) | 9.677 (33.7) | 16.94 (46.6) | 31.72 (11.4)
  Nor-S-297995 Day 1 (n = 9, 8, 7) | NA (NA) — Not calculable as plasma concentrations of Nor-S-297995 on Day 1 were below the limit of quantification. | 0.5106 (55.5) | 2.950 (53.8)
  Nor-S-297995 Day 28 (n = 3, 4, 3) | 0.3522 (896.9) | 0.8158 (463.1) | 2.256 (140.0)

36. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse events (TEAEs) were adverse events that occurred after the first dose of study drug.
  Treatment-related TEAEs were defined as TEAEs that were considered by the Investigator to be definitely, probably, or possibly related to study drug.
Time Frame: From first dose of study drug through 28 days after the last dose of study treatment (up to 57 days).
Population: Adverse events were assessed using the safety population. The safety population included all participants who received study drug. This population was analyzed as treated.
Measure: Number; unit: participants
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Number analyzed (Participants) | 61 | 61 | 60 | 61
participants
  TEAEs | 31 | 25 | 30 | 34
  Treatment-related TEAEs | 10 | 10 | 15 | 24
  Serious TEAEs | 0 | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 28 days after the last dose of study treatment (up to 57 days).
Description: The safety population included all participants who received study drug.
Arm/Group | Placebo | Naldemedine 0.1 mg | Naldemedine 0.2 mg | Naldemedine 0.4 mg
Serious Adverse Events (participants affected / at risk) | 0/61 | 2/61 | 0/60 | 1/61
Other Adverse Events (participants affected / at risk) | 19/61 | 15/61 | 19/60 | 28/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=61) | Naldemedine 0.1 mg (N=61) | Naldemedine 0.2 mg (N=60) | Naldemedine 0.4 mg (N=61)
Chest pain (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1
Appendicitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=61) | Naldemedine 0.1 mg (N=61) | Naldemedine 0.2 mg (N=60) | Naldemedine 0.4 mg (N=61)
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 5 | 9
Diarrhea (Gastrointestinal disorders) | 3 | 3 | 3 | 11
Flatulence (Gastrointestinal disorders) | 2 | 3 | 3 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Anorectal discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 3 | 4
Influenza (Infections and infestations) | 2 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 1
Influenza like illness (General disorders) | 0 | 2 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 1 | 2 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Hot flush (Vascular disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.